CLINICAL TRIAL: NCT04572620
Title: Retrospective Chart Review of Children With Primary Immunodeficiencies (PID) Who Received Targeted Therapy of Interstitial Lymphocytic Lung Disease (ILLD) With Abatacept or Rituximab.
Brief Title: Rituximab and Abatacept Effectiveness in Differential Treatment of Interstitial Lymphocytic Lung Disease in Children With Primary Immunodeficiencies.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: NCPHOI-2020-08
Record Dates: First submitted 2020-09-21; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Interstitial Lymphocytic Lung Disease
Keywords: interstitial lymphocytic lung disease; primary immunodeficiency; children; treatment; rituximab; abatacept
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Rituximab; Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1(rituximab)
  Interventions: Drug: Rituximab
- group 2 (abatacept)
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 as 4 weekly consecutive i.v. infusions with subsequent infusions of 375 mg/m2 performed every 3 months for 12 months.
  Groups: group 1(rituximab)
Drug: Abatacept — 10 mg/kg i.v. every 2 weeks twice, then every 4 weeks for 12 months.
  Groups: group 2 (abatacept)

SUMMARY:
The rationale for this retrospective study is to evaluate the efficacy and safety of abatacept and rituximab treatment of ILLD in a cohort of pediatric patients with different forms of PID, who received one of the two therapy regimens predominantly based on the lesions histopathology.

DETAILED DESCRIPTION:
Primary immunodeficiencies (PID) represent a heterogeneous group of more than 400 inherited conditions with associated immune dysfunctions. Though severe recurrent/chronic infections are the main cause of mortality and morbidity in PID, immune dysregulation manifesting with oncological and autoimmune or autoinflammatory conditions involving various organs and systems have been the focus of research in the recent years.

The interstitial lymphocytic lung disease (ILLD) is one of the recently characterized non-malignant PID complications. Immune dysregulation in ILLD causes reactive bronchi-associated lymphoid tissue (BALT) hyperplasia that manifests in several pathomorphological forms: follicular bronchiolitis (FB), nodular lymphoid hyperplasia (NLH), and lymphocytic interstitial pneumonia (LIP). Treatment of ILLD patients with various immunosuppressive drugs leads to inconsistent results ranging from partial\transient effect to no effect at all and has been often associated with adverse effects and an increase in infections' rate. Therefore there is a need for targeted therapy of ILLD. In small cohorts of adult PID patients rituximab in combination with azathioprine proved to be effective. Yet, the reports are scarce and there is currently no consensus on ILLD treatment, especially in children.

The study will collect and analyze information on the effectiveness and safety of ILLD monotherapy with rituximab or abatacept, chosen predominantly based on the pathomorphological characteristics of lymphoid infiltration, as well as genetic defects, in a cohort of pediatric patients with PID.

ELIGIBILITY:
Inclusion Criteria:

1. Histological and/or radiological diagnosis of ILLD.
2. Treatment with rituximab or abatacept for at least 12 months.
3. No signs of ongoing infectious pulmonary process at the start of the treatment.
4. Regular IG substitution with trough IgG levels > 5g/l.

Exclusion criteria are nonadherence to therapy.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with interstitial lymphocytic lung disease treated in Dmitry Rogachev National Research and Clinical Center for Pediatric Hematology, Oncology and Immunology, Moscow, Russia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Dynamics of severity clinical and radiological symptoms | before the time the first dose of study treatment was administered
  Dynamics of severity clinical and radiological symptoms of ILLD using scale score.
Dynamics of severity clinical and radiological symptoms | 3 months of treatment
  Dynamics of severity clinical and radiological symptoms of ILLD using scale score.
Dynamics of severity clinical and radiological symptoms | 6 months of treatment
  Dynamics of severity clinical and radiological symptoms of ILLD using scale score.
Dynamics of severity clinical and radiological symptoms | 1 year of treatment
  Dynamics of severity clinical and radiological symptoms of ILLD using scale score.

SECONDARY OUTCOMES:
Frequency of adverse events | from the time the first dose of study treatment was administered until 12 mo of treatment
quality of life of patients | before the time the first dose of study treatment was administered until 12 mo of treatment
  The quality of life of patients before and after therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Research and Clinical Center for Pediatric Hematology, Oncology and Immunology, Moscow, Russia